CLINICAL TRIAL: NCT00794664
Title: A Prospective Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of Mipomersen in Patients With Severe Hypercholesterolemia on a Maximally Tolerated Lipid-Lowering Regimen and Who Are Not on Apheresis
Brief Title: Safety and Efficacy of Mipomersen in Patients With Severe Hypercholesterolemia on a Maximally Tolerated Lipid-Lowering Regimen and Who Are Not on Apheresis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIPO3500108; 2008-006020-53 (EudraCT Number)
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Results first posted 2013-03-21 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-08

CONDITIONS: Hypercholesterolemia; Coronary Heart Disease
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease | interventions — mipomersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Weekly subcutaneous injections for 26 weeks
  Interventions: Drug: Placebo
- Mipomersen (Experimental): 200 mg weekly subcutaneous injections for 26 weeks
  Interventions: Drug: Mipomersen

INTERVENTIONS:
Drug: Mipomersen — 200 mg (1 mL), weekly subcutaneous injections for 26 weeks
  Other Names: ISIS 301012; Mipomersen sodium; Kynamro™
  Arms: Mipomersen
Drug: Placebo — 1 mL weekly subcutaneous injections for 26 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of dosing with mipomersen for 26 weeks in treating severely hypercholesterolemic patients who are on a maximally tolerated lipid-lowering regimen and who are not on apheresis.

DETAILED DESCRIPTION:
Hypercholesterolemia is characterized by markedly elevated low density lipoproteins (LDL). Elevated LDL is a major risk factor for coronary heart disease (CHD).

Mipomersen is an antisense drug that reduces a protein in the liver cells called apolipoprotein B (Apo-B). Apo-B plays a role in producing low density lipoprotein cholesterol (LDL-C) (the "bad" cholesterol) and moving it from the liver to one's bloodstream. High LDL-C is an independent risk factor for the development of coronary heart disease (CHD) or other diseases of blood vessels. It has been shown that lowering LDL-C reduces the risk of heart attacks and other major adverse cardiovascular events. The purpose of this study is to determine whether mipomersen safely and effectively lowers LDL-C in severely hypercholesterolemic patients who are on a maximally tolerated lipid-lowering regimen and who are not on apheresis.

ELIGIBILITY:
Inclusion Criteria:

* Fasting LDL-C ≥200 mg/dL (5.1 mmol/L) at screening and the presence of at least 1 of the following criteria:

  * Myocardial infarction (MI)
  * Percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)
  * Coronary artery disease documented by angiography or any other accepted imaging technique
  * Positive exercise test (≥1 mm ST-depression at maximal exercise or test terminated because of angina) or a perfusion defect (e.g., thallium or single photon emission computed tomography)
  * Other clinical atherosclerotic diseases: peripheral artery disease, symptomatic carotid artery disease, abdominal aortic aneurysm
  * Or, if alternative above were not met, fasting LDL-C ≥300 mg/dL (7.8 mmol/L)
* On stable, maximally tolerated statin therapy for 8 weeks
* On stable, medication from an additional class of hypolipidemic agents for 8 weeks.
* On stable, low fat diet for 12 weeks
* Stable weight for 6 weeks

Exclusion Criteria:

* Significant health problems in the recent past including heart attack, stroke, coronary syndrome, unstable angina, heart failure, significant arrhythmia, hypertension, blood disorders, liver disease, cancer, digestive disorders, Type I diabetes, or uncontrolled Type II diabetes
* Apheresis within 3 months prior to Screening or expected to start apheresis during the treatment phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (26):
- United States (9):
  - Jupiter, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Kansas City, Kansas
  - Boston, Massachusetts
  - St Louis, Missouri
  - Concord, New Hampshire
  - Cincinnati, Ohio
  - Aiken, South Carolina
- Canada (3):
  - Winnipeg, Manitoba
  - Chicoutimi, Quebec
  - Montreal, Quebec
- Czechia (4):
  - Hardec Kralove
  - Pilsen
  - Prague
  - Uherské Hradiště
- Germany (4):
  - Berlin
  - Freiburg im Breisgau
  - Heidelberg
  - Koln (Lindenthal)
- South Africa (3):
  - Cape Town
  - Gauteng
  - Pretoria
- United Kingdom (3):
  - Guildford, Surrey
  - London
  - Manchester

REFERENCES:
- [Result] McGowan MP, Tardif JC, Ceska R, Burgess LJ, Soran H, Gouni-Berthold I, Wagener G, Chasan-Taber S. Randomized, placebo-controlled trial of mipomersen in patients with severe hypercholesterolemia receiving maximally tolerated lipid-lowering therapy. PLoS One. 2012;7(11):e49006. doi: 10.1371/journal.pone.0049006. Epub 2012 Nov 13. PMID 23152839
- [Derived] Duell PB, Santos RD, Kirwan BA, Witztum JL, Tsimikas S, Kastelein JJP. Long-term mipomersen treatment is associated with a reduction in cardiovascular events in patients with familial hypercholesterolemia. J Clin Lipidol. 2016 Jul-Aug;10(4):1011-1021. doi: 10.1016/j.jacl.2016.04.013. Epub 2016 May 9. PMID 27578134
- [Derived] Santos RD, Raal FJ, Catapano AL, Witztum JL, Steinhagen-Thiessen E, Tsimikas S. Mipomersen, an antisense oligonucleotide to apolipoprotein B-100, reduces lipoprotein(a) in various populations with hypercholesterolemia: results of 4 phase III trials. Arterioscler Thromb Vasc Biol. 2015 Mar;35(3):689-99. doi: 10.1161/ATVBAHA.114.304549. Epub 2015 Jan 22. PMID 25614280

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One hundred and four patients were screened and 58 randomized in a 2:1 treatment arm ratio.
Period: Treatment Period
Arm/Group | Placebo | Mipomersen
Started | 19 | 39
Completed | 18 (3 participants enrolled in open-label extension study NCT00694109) | 27 (6 participants enrolled in open-label extension study NCT00694109)
Not Completed | 1 | 12
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol non-compliance | 0 | 1
Not completed — Other | 0 | 1
Not completed — Adverse Event | 1 | 8
Period: Follow-up Period
Arm/Group | Placebo | Mipomersen
Started | 16 (Participants enrolled in the open-label extension (NCT00694109) or continued in the follow-up period) | 33 (Participants enrolled in the open-label extension (NCT00694109) or continued in the follow-up period)
Completed | 15 | 28
Not Completed | 1 | 5
Not completed — Other | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mipomersen | Total
Number analyzed (Participants) | 19 | 39 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (13.5) | 51.8 (14.3) | 50.5 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 21 | 33
  Male | 7 | 18 | 25
Race/Ethnicity, Customized [Number; unit: participants]
  White | 16 | 33 | 49
  Black | 1 | 2 | 3
  Asian | 0 | 1 | 1
  Multiple | 2 | 1 | 3
  Other | 0 | 2 | 2
Ethnicity [Number; unit: participants]
  Not Hispanic or Latino | 19 | 39 | 58
  Hispanic or Latino | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.9 (4.10) | 28.4 (5.35) | 28.9 (4.98)
Waist/hip ratio [Mean (Standard Deviation); unit: ratio] | 0.94 (0.06) | 0.92 (0.09) | 0.93 (0.08)
Metabolic syndrome [Number; unit: participants] — Yes if 3 or more risk factors are present: 1) Abdominal obesity 2) Triglycerides >=150 mg/dl * 3) High density lipoprotein cholesterol (men <40 mg/dl) (women <50 mg/dl) * 4) Systolic blood pressure >=130 or diastolic >=85 mmHg * 5) Fasting glucose >=100 mg/dl * * = or on medication for condition
  participants
    No | 10 | 25 | 35
    Yes | 9 | 14 | 23
Tobacco Use [Number; unit: participants]
  Current | 5 | 4 | 9
  Non-current | 7 | 11 | 18
  Never | 7 | 24 | 31
Alcohol Use [Number; unit: participants]
  Current | 7 | 27 | 34
  Non-current | 4 | 5 | 9
  Never | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at Primary Efficacy Time Point
Description: LDL-C was measured in mg/dL. Samples were taken following an overnight fast. For patients with triglycerides <400 mg/dL, LDL-C was obtained using Friedewald's calculation; and for patients with triglycerides >=400 mg/dL, LDL-C was directly measured by the central laboratory using ultracentrifugation. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: Baseline (the average of the screening and Day 1 pre-treatment assessments) and the Primary Efficacy Time point (PET) up to week 28
Population: Full analysis set (FAS). The FAS, which represents the practically-feasible intent-to-treat (ITT) population as delineated in ICH Guideline E9, consists of treated participants with a valid baseline and at least one post-baseline LDL-C measure.
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
percentage of baseline | 12.5 (46.87) | -35.9 (24.71)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Based upon prior clinical study experience with mipomersen, it was estimated that the standard deviation of the percent change in LDL-C was approximately 22%. With 15 patients in the control group and 30 patients in the mipomersen-treated group, this study would have at least 80% power to detect a 20 percentage point difference between the 2 treatment groups. Enrollment was to be conducted such that at least 51 patients were randomized to allow for potential exclusions from an analysis set; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Statistical significance was concluded if p≤0.05

2. Primary Outcome: LDL-C at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
mg/dL
  Baseline | 249.4 (84.3) | 276.1 (72.1)
  PET | 263.9 (102.0) | 174.9 (82.8)

3. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo-B) at Primary Efficacy Time Point
Description: Apo-B was measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
percentage of baseline | 11.41 (36.80) | -35.88 (22.95)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Inflation of type 1 error was controlled by specifying a small number of secondary parameters and a sequential inferential approach in which inferential conclusions about each successive parameter required statistical significance of the prior one

4. Secondary Outcome: Apo-B at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
mg/dL
  Baseline | 182.8 (48.6) | 202.1 (49.1)
  PET | 193.7 (54.2) | 126.8 (49.6)

5. Secondary Outcome: Percentage Change From Baseline in Total Cholesterol at Primary Efficacy Time Point (PET)
Description: Total cholesterol was measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
percentage of baseline | 11.13 (34.74) | -28.31 (20.43)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Inferential conclusions about this parameter require statistical significance of the previous secondary outcome measure (i.e., percent change from baseline in Apo B at PET)

6. Secondary Outcome: Total Cholesterol at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
mg/dL
  Baseline | 320.6 (87.2) | 356.8 (77.0)
  PET | 341.5 (100.5) | 251.5 (82.2)

7. Secondary Outcome: Percentage Change From Baseline in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) at Primary Efficacy Time Point (PET)
Description: Non-HDL-C was measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
percentage of baseline | 14.17 (47.75) | -33.95 (23.80)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Inferential conclusions about this parameter require statistical significance of the previous secondary outcome measure (i.e., percent change from baseline in total cholesterol at PET)

8. Secondary Outcome: Non-HDL-C at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
mg/dL
  Baseline | 277.5 (88.3) | 305.6 (78.3)
  PET | 296.7 (103.8) | 198.1 (85.3)

9. Other Pre Specified Outcome: Percentage Change From Baseline in Triglycerides at Primary Efficacy Time Point (PET)
Description: Triglycerides were measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
percentage of baseline | 26.50 (60.61) | -8.71 (40.10)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.034, t-test, 2 sided — Statistical significance was concluded if p ≤0.05

10. Other Pre Specified Outcome: Triglycerides at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
mg/dL
  Baseline | 140.3 (49.8) | 142.2 (86.0)
  PET | 164.5 (61.2) | 116.3 (63.3)

11. Other Pre Specified Outcome: Percentage Change From Baseline in Lipoprotein(a) at Primary Efficacy Time Point (PET)
Description: Lipoprotein(a) was measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
percentage of baseline | -1.46 (25.74) | -32.65 (32.98)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Statistical significance was concluded if p ≤0.05

12. Other Pre Specified Outcome: Lipoprotein(a) at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
mg/dL
  Baseline | 32.4 (28.5) | 61.3 (68.4)
  PET | 32.1 (28.1) | 43.3 (54.3)

13. Other Pre Specified Outcome: Percentage Change From Baseline in Very-Low-Density Lipoprotein Cholesterol (VLDL-C) at Primary Efficacy Time Point (PET)
Description: VLDL-C was measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
percentage of baseline | 25.13 (58.66) | -9.36 (39.57)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.032, t-test, 2 sided — Statistical significance was concluded if p ≤0.05

14. Other Pre Specified Outcome: VLDL-C at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
mg/dL
  Baseline | 28.1 (9.9) | 29.1 (20.0)
  PET | 32.8 (12.3) | 23.2 (12.6)

15. Other Pre Specified Outcome: Change From Baseline in Ratio of Low-density Lipoprotein Cholesterol (LDL-C) to High-density Lipoprotein Cholesterol (HDL-C) at Primary Efficacy Time Point (PET)
Description: LDL-C and HDL-C were measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
percentage of baseline | 1.9 [-14.3 to 18.0] | -41.8 [-57.4 to -16.4]
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p < 0.001, Wilcoxon rank sum test — Statistical significance was concluded if p ≤0.05

16. Other Pre Specified Outcome: Ratio of LDL-C to HDL-C at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
ratio
  Baseline | 5.89 [3.89 to 6.58] | 5.21 [4.13 to 6.97]
  PET | 5.85 [3.28 to 7.76] | 3.05 [2.11 to 4.26]

17. Other Pre Specified Outcome: Percent Change From Baseline in Apolipoprotein A1 (Apo-A1) at Primary Efficacy Time Point (PET)
Description: Apo-A1 was measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
percentage of baseline | 1.75 (14.33) | -3.04 (15.76)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.278, t-test, 2 sided — Statistical significance was concluded if p ≤0.05

18. Other Pre Specified Outcome: Apo-A1 at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
mg/dL
  Baseline | 139.2 (32.6) | 154.9 (31.4)
  PET | 140.7 (34.2) | 147.9 (27.0)

19. Other Pre Specified Outcome: Percentage Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C) at Primary Efficacy Time Point (PET)
Description: HDL-C was measured in mg/dL. Samples were taken following an overnight fast. Baseline was defined as the average of the screening and Study Day 1 (pre-treatment) assessments. An assessment was not included in this calculation if it was associated with a non-fasting blood draw or was drawn more than 4 weeks prior to Study Day 1. The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
percentage of baseline | 3.16 (16.50) | 5.78 (21.25)
Statistical Analysis 1: Comparison: Placebo vs Mipomersen; Test type: Superiority or Other; p = 0.647, t-test, 2 sided — Statistical significance was concluded if p ≤0.05

20. Other Pre Specified Outcome: HDL-C at Baseline and the Primary Efficacy Time Point (PET)
Description: The PET was the post-baseline visit, for which LDL-C was assessed, closest to 14 days after the last dose of study drug.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Mipomersen
Number analyzed (Participants) | 18 | 39
mg/dL
  Baseline | 43.1 (11.6) | 51.1 (15.1)
  PET | 44.8 (16.3) | 53.4 (16.7)

ADVERSE EVENTS:
Time Frame: Day 1 to week 28. On-treatment AEs started on/after the first study drug dose and on/before the end of the treatment period. The treatment period was the time study drug was administered until the later of the PET or 14 days after last study drug dose.
Description: The Safety Set includes all randomized patients who receive at least 1 injection of the study treatment. In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Placebo | Mipomersen
Serious Adverse Events (participants affected / at risk) | 0/19 | 6/39
Other Adverse Events (participants affected / at risk) | 16/19 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | Mipomersen (N=39)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 1
Device malfunction (General disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | Mipomersen (N=39)
Angina pectoris (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Eye swelling (Eye disorders) | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 5
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 4
Influenza like illness (General disorders) | 0 | 9
Injection site discolouration (General disorders) | 0 | 3
Injection site erythema (General disorders) | 2 | 22
Injection site haematoma (General disorders) | 4 | 9
Injection site induration (General disorders) | 0 | 3
Injection site inflammation (General disorders) | 0 | 3
Injection site mass (General disorders) | 0 | 1
Injection site nodule (General disorders) | 0 | 1
Injection site oedema (General disorders) | 0 | 5
Injection site pain (General disorders) | 0 | 23
Injection site papule (General disorders) | 0 | 1
Injection site pruritus (General disorders) | 1 | 13
Injection site rash (General disorders) | 0 | 3
Injection site reaction (General disorders) | 0 | 2
Injection site recall reaction (General disorders) | 0 | 2
Injection site swelling (General disorders) | 0 | 12
Injection site urticaria (General disorders) | 0 | 1
Injection site vesicles (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 4
Liver tenderness (Hepatobiliary disorders) | 0 | 1
Allergy to plants (Immune system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 4
Onychomycosis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pleurisy viral (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 3
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 7
Aspartate aminotransferase increased (Investigations) | 0 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 0 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 2
Cardiac murmur (Investigations) | 0 | 1
Electrocardiogram PR prolongation (Investigations) | 0 | 1
Epstein-Barr virus antibody positive (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 1
Lethargy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 2
Renal cyst (Renal and urinary disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Xanthoma (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 3
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish site data after a multi-centered publication or 12 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 6 months (contracts have variable timeframes) upon notifying PI that it will file a patent application on inventions contained in the draft.